CLINICAL TRIAL: NCT00497692
Title: Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability and Dermical Sensitivity) for Dermacyd Femina Delicata
Brief Title: Topic Compatibility Lactoserum (Dermacyd Delicata - New Fragrance)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACTO_L_02948
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactoserum

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd Femina Delicata.

ELIGIBILITY:
Inclusion Criteria:

* Phototypes: I, II, III and IV
* Integral skin test in the region

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Use of antinflammatory or immune-suppression drugs
* Personal history of atopy
* History of sensibilization or irritation for topic products
* Active cutaneous disease
* Use of new drugs and/or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Score evaluation of the cutaneous reaction, preconized by International Contact Dermatitis Research Group (ICDRG) | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, São Paulo, Brazil